CLINICAL TRIAL: NCT07224763
Title: EXTEND: A Prospective Study to Evaluate the Safety and Efficacy of GGTA1 KO Thymokidney XenoTransplantation in Patients With End-stage Renal Disease (ESRD)
Brief Title: Study to Evaluate the Safety and Efficacy of the GGTA1 KO Thymokidney in Patients With ESRD
Acronym: EXTEND
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GPT-KF-101
Record Dates: First submitted 2025-11-04; First posted 2025-11-05 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: ESRD (End-Stage Renal Disease); Kidney Transplantation; Xenotransplantation
Keywords: End-stage renal disease; ESRD; Xenotransplantation; GGTA1 KO Thymokidney
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: This single group study will enroll participants simultaneously from either of 2 patient populations: (1) participants that are ineligible for conventional allogeneic kidney transplantation due to medical reason(s) or (2) participants on an OPTN kidney transplant waitlist that are more likely to die or go untransplanted within 5 years than receive a kidney transplant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GGTA1 KO Thymokidney (Experimental): Participants will receive GGTA1 KO Thymokidney
  Interventions: Biological: GGTA1 KO Thymokidney

INTERVENTIONS:
Biological: GGTA1 KO Thymokidney — Porcine kidney containing an intentional genomic alteration and thymic tissue autograft for xenotransplantation

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the GGTA1 KO Thymokidney in patients with end-stage renal disease (ESRD) who are either not eligible for conventional allogeneic kidney transplantation (Group 1) or are on an Organ Procurement and Transplantation Network (OPTN) kidney transplant waitlist, but are more likely to die or go untransplanted within 5 years than receive a kidney transplant (Group 2).

The study consists of xenotransplantation followed by a 24-week Post-transplant Follow-up Period (Part A) to evaluate the efficacy and safety objectives followed by a Long-term Follow-up Period (Part B) to evaluate participant survival, GGTA1 KO Thymokidney survival, and screening for zoonotic infections. Part B will continue for the lifetime of the participant or for 52 weeks following nephrectomy, if required.

DETAILED DESCRIPTION:
This is a Phase 1/2/3, multicenter, open-label, safety and efficacy study of the GGTA1 KO Thymokidney in patients with ESRD. The study will be comprised of the following:

* A Screening Period up to 52 weeks.
* Part A consists of the GGTA1 KO Thymokidney transplantation followed by a 24-week Post-transplant Follow-up Period, including the evaluation of all study endpoints and safety assessments.
* Part B is a Long-term Follow-up Period that extends for the lifetime of participants who received the GGTA1 KO Thymokidney or for 52 weeks following nephrectomy, if required, including but not limited to documentation of participant survival, GGTA1 KO Thymokidney survival, and screening for zoonotic infections.

There will be 2 groups of participants enrolled in the study. Group 1 will be participants deemed ineligible for conventional allogeneic kidney transplantation due to medical reason(s). Group 2 will be participants on an OPTN kidney transplant waitlist but who are more likely to die or go untransplanted within 5 years than receive a kidney transplant.

For the purpose of the primary analysis, the end of the study is defined as the date of the final visit of the final participant in Part A of the study.

ELIGIBILITY:
Inclusion Criteria for all Participants (Groups 1 and 2):

1. Provide voluntarily informed consent to participate in the study and for lifetime follow-up.
2. Have a diagnosis of ESRD at the time of informed consent.
3. Hemodialysis dependent for a minimum of 6 months and has a functioning arterial-venous fistula/graft or permanent catheter at the time of informed consent.
4. 50 to 70 years of age at the time of informed consent, or 40 to <50 years of age with a calculated panel reactive antibody (cPRA) of ≥99.9%.
5. Evidence of thymic involution on chest computed tomography (CT) scan with a thymic region of interest score of ≤1.
6. Live within 3 hours travel time of the xenotransplant center.
7. Female participants must be postmenopausal or permanently sterilized (eg, hysterectomy, bilateral oophorectomy, or bilateral salpingectomy). Male participants must agree to the use of a highly effective method of birth control, if the possibility of conception exists.
8. Negative xeno-crossmatch at Screening and pre-transplant.
9. Estimated Post Transplant Survival Calculator score >20%.(https://optn.transplant.hrsa.gov/data/allocation-calculators/epts-calculator/).
10. Body mass index ≤35 kg/m2.
11. Have completed or have initiated and plan to complete (meningococcal A, C, W, Y and meningococcal B vaccine series only) Centers for Disease Control and Prevention-recommended courses of age- and risk-factor-appropriate vaccinations.
12. Seropositive (immunoglobulin G) for cytomegalovirus and Epstein-Barr virus.

Additional Inclusion Criteria for Group 1:

1. Ineligible for conventional allogeneic kidney transplantation due to medical reason(s) for any of the following:

1. Ineligible for a living donor transplant.
2. Ineligible for an OPTN kidney transplant waitlist (reason for ineligibility will be collected).
3. Delisted from OPTN kidney transplant waitlist (reason for delisting will be collected).

Additional Inclusion Criteria for Group 2:

1. On an OPTN kidney transplant waitlist (active or inactive status).
2. No approved living kidney donors.
3. More likely to die or go untransplanted within 5 years than receive a kidney transplant as measured by the Kidney Transplant Decision Aid at the time of informed consent (select United States for "Choose your state" field and National average for "Choose your transplant program" field; https://www.srtr.org/tools/kidney-transplant-decision-aid/).

Exclusion Criteria (pertain to all participants in Groups 1 and 2):

1. Need for multiple organ transplants.
2. Severe medical co-morbidities including, but not limited to:

   1. Chronic liver disease.
   2. Advanced cardiovascular disease.
   3. Severe peripheral vascular disease that limits technical ability to transplant the GGTA1 KO Thymokidney.
   4. Severe neurologic diseases or conditions that would preclude meaningful recovery or informed consent.
   5. Oral steroid-dependent airway disorder or chronic pulmonary disease or requires chronic, intermittent, or continuous supplemental oxygen.
   6. Pulmonary hypertension.
   7. Uncontrolled diabetes or sequelae of diabetes mellitus including severe non-proliferative diabetic retinopathy.
   8. Severe neurogenic bladder that requires intermittent catheterization.
3. ESRD due to hereditary or structural kidney disease.
4. Active or recently treated malignancy at the time of informed consent.
5. Non-renal cause of hematological disorders associated with anemia (eg, thalassemia and sickle disease).
6. Cannot discontinue chronic anticoagulation therapy (low-dose daily aspirin is permissible).
7. History of major psychiatric disorders with psychiatric hospitalization and/or suicidal ideation within 5 years of informed consent.
8. Being treated for active tuberculosis (TB), have received prophylaxis for positive FDA-approved interferon-gamma release assay, or test positive for TB by FDA-approved interferon-gamma release assay test during Screening.
9. Nucleic acid test (NAT) positive for hepatitis B virus and/or hepatitis C virus, hepatitis B surface antibody (anti-HBs) titer <10 mIU/mL unless the participant is determined to be a nonresponder to hepatitis B vaccination (a nonresponder is defined as having an anti-HB titer <10 mIU/mL after having completed both the standard vaccine series and a fourth booster dose and/or second standard vaccine series), and/or positive for human immunodeficiency virus (HIV; HIV-1 and HIV-2 antibody and/or NAT).
10. Not able to independently perform activities of daily life.
11. Have a history of medical noncompliance that may preclude adherence to the demands and requirements of xenotransplantation (eg, history of substance use disorder [SUD] within 1 year of informed consent, lack of social support, untreated psychological conditions).

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2076-03 (Estimated)

PRIMARY OUTCOMES:
Survival Rate of Patients with ESRD Receiving the GGTA1 KO Thymokidney at 24 Weeks Post Transplant | Day 0 (day of xenotransplantation) to 24 weeks post transplant
  Participant survival rate at 24 weeks post transplant.
Survival Rate of the GGTA1 KO Thymokidney at 24 Weeks Post Transplant | Day 0 (day of xenotransplantation) to 24 weeks post transplant
  GGTA1 KO Thymokidney survival rate at 24 weeks post transplant. GGTA1 KO Thymokidney failure is defined as GGTA1 KO Thymokidney nephrectomy.
Survival Time of Participants Receiving the GGTA1 KO Thymokidney | Day 0 (day of xenotransplantation) until death for any cause, assessed at least every 24 weeks after transplantation while the participant is alive, up to 50 years
  Participant survival post transplant. Participant survival is defined as time from xenotransplantation to death for any cause.
Survival Time of the GGTA1 KO Thymokidney (Overall Survival) | Day 0 (day of xenotransplantation) until start of chronic dialysis, nephrectomy, or death, whichever occurs first, assessed at least every 24 weeks after transplantation while the participant is alive and the thymokidney is functional, up to 50 years
  Overall survival of the GGTA1 KO Thymokidney post transplant. Overall survival time of the GGTA1 KO Thymokidney is defined as time from xenotransplantation to GGTA1 KO Thymokidney nephrectomy or death, whichever occurs first.
Survival Time of the GGTA1 KO Thymokidney (Death-censored Survival) | Day 0 (day of xenotransplantation) until start of chronic dialysis, nephrectomy, or death, whichever occurs first, assessed at least every 24 weeks after transplantation while the participant is alive and the thymokidney is functional, up to 50 years
  Death-censored survival GGTA1 KO Thymokidney. Death-censored survival time of the GGTA1 KO Thymokidney is defined as time from xenotransplantation to GGTA1 KO Thymokidney nephrectomy censored for death.
GGTA1 KO Thymokidney Function Post Transplant (Endogenous GFR) | At 24 weeks post transplant
  Endogenous measured GFR (24-hour urine creatinine clearance) at 24 weeks post transplant.
GGTA1 KO Thymokidney Function Post Transplant (Exogenous GFR) | At 24 weeks post transplant
  Exogenous measured GFR (nuclear medicine GFR) at 24 weeks post transplant.
GGTA1 KO Thymokidney Function Post Transplant (Proliferative Responsiveness) | At 24 weeks post transplant
  Proliferative responsiveness to source GGTA1 KO Pig versus third-party pig as measured by mixed lymphocyte reaction from baseline to 24 weeks post transplant.
Quality of Life in Participants Receiving the GGTA1 KO Thymokidney by EuroQol 5-Dimension 5-Level (EQ-5D-5L) | Baseline to 24 weeks post transplant
  Change in the EQ-5D-5L from baseline to 24 weeks post transplant. The EQ-5D-5L questionnaire assesses health-related quality of life across 5 categories (Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression).
  Each category has 5 levels, ranging from 1 (no problems) to 5 (extreme problems or inability to perform the activity). Higher scores indicate a worse health outcome (more mobility issues, greater pain, more anxiety, etc).
Quality of Life in Participants Receiving the GGTA1 KO Thymokidney by Standardized Outcomes in Nephrology Life Participant (SONG-LP) | Baseline to 24 weeks post transplant
  Change in SONG-LP from baseline to 24 weeks post transplant. The SONG-LP assesses participation in different life activities over the past month. The minimum score (worst outcome) is 4 (if all responses are "1" - Never) and the maximum score (best outcome) is 20 (if all responses are "5" - Always). Higher scores indicate a better health outcome (greater ability to participate in activities).
Quality of Life in Participants Receiving the GGTA1 KO Thymokidney by Kidney Transplant Questionnaire (KTQ) | Baseline to 24 weeks post transplant
  Change in KTQ from baseline to 24 weeks post transplant. Each question in the KTQ is scored on a 1 to 7 scale with: 1 = worst outcome (eg, "A very great deal of trouble or distress" / "All of the time") and 7 = best outcome (eg, "No trouble or distress" / "None of the time"). Higher scores indicate a better outcome, meaning less distress, fewer symptoms, and better well-being.
Quality of Life in Participants Receiving the GGTA1 KO Thymokidney by Patient Global Impression of Change (PGI-C) | At 24 weeks post transplant
  PGI-C at 24 weeks post transplant. The PGI-C assesses a patient's perception of improvement or worsening over time. The minimum score (best outcome) is 1 ("Very Much Improved") and the maximum score (worst outcome) is 7 ("Very Much Worse"). Higher scores indicate a worse health outcome (greater worsening).
Incidence of Treatment-Emergent Adverse Events (Safety of the GGTA1 KO Thymokidney) | Baseline until last visit, assessed at least every 24 weeks after transplantation while the participant is alive and the thymokidney is functional, up to 50 years, or for 1 year after nephrectomy if required
  Incidence of adverse events and serious adverse events; all-cause mortality.
Incidence of Proteinuria | Day 0 (day of xenotransplantation) until last visit, assessed at least every 24 weeks after transplantation while the participant is alive and the thymokidney is functional, up to 50 years, or for 1 year after nephrectomy if required
  Incidence of proteinuria from Day 0.
Incidence of Zoonotic Infection | Day 0 (day of xenotransplantation) until last visit, assessed at least every 24 weeks after transplantation while the participant is alive and the thymokidney is functional, up to 50 years, or for 1 year after nephrectomy if required
  Incidence of zoonotic infection from Day 0.
Incidence of Opportunistic Infection | Day 0 (day of xenotransplantation) until last visit, assessed at least every 24 weeks after transplantation while the participant is alive and the thymokidney is functional, up to 50 years, or for 1 year after nephrectomy if required
  Incidence of opportunistic infection from Day 0.

CONTACTS AND LOCATIONS:
Locations (1):
- New York University Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No